CLINICAL TRIAL: NCT02880774
Title: Influence of Manual Therapy in Temporomandibular Joint on the Mandibular Movement: Clinical Trial, Randomised, Placebo-controlled and Blind
Brief Title: Influence of Manual Therapy in Temporomandibular Joint Disorder
Acronym: THERAPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Daniela Aparecida Biasotto-Gonzalez, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uninove_Reabilitação
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Musculoskeletal Diseases
Keywords: Temporomandibular Joint Disorders; Mandibular Movement; Músculoesqueléticas Manipulations; Modalities of Physiotherapy.
MeSH Terms: conditions — Musculoskeletal Diseases; Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mandibular Nonspecific mobilization (Experimental): GA: Mandibular Nonspecific mobilization on the region of the face with presence of TMD.
  Interventions: Other: mandibular nonspecific mobilization
- ultrasound detuned (Placebo Comparator): Group B: Used ultrasound equipment detuned on the region of the face with presence of TMD.
  Interventions: Other: Ultrasound detuned,

INTERVENTIONS:
Other: mandibular nonspecific mobilization — The mobilization will be held with the individual in supine position, by a trained and experienced therapist, where using disposable gloves, will position the first finger on the last molar, performing intermittently mobilization during 1 minute, will be held five repetitions. Going on a break during the repetition, in that the individual will carry out 15 times language exercises on the palate. With regard to mobilizing joint side, this will be previously set by means of the RDC/TMD and may be unilateral or bilateral basis, depending on the diagnosis. The therapist will remain in orthostatic in opposite side the mobilization to prevent any pressure on the jaw. The treatment will last for 4 weeks, 3 times a week, for a total of 12 sessions.
  Other Names: mandibular mobilization
  Arms: Mandibular Nonspecific mobilization
Other: Ultrasound detuned, — Will be held the identical positioning to group A with the individual supine on the stretcher, used ultrasound equipment detuned on the region of the face with the presence of TMD. The procedures of this group will have a duration of 4 weeks, 3 times a week, for a total of 12 sessions.
  Arms: ultrasound detuned

SUMMARY:
Introduction: Temporomandibular joint dysfunction (TMD) is characterized for being a complex and multifactorial pathology, where functional and pathological changes commit temporomandibuar articulation, masticatory muscles, and other associated structures. In the light of the whole complexity of the DTM noted the necessity of interdisciplinary treatment, including physical therapy with the use of manual features, has been excelling. Objective: The aim of this study is to evaluate the influence of mandibular nonspecific mobilization on the mandibular movement and lateralidades, through the three-dimensional kinematics in subjects with diagnosis of TMD, as well as analyze the behavior of pain, quality of life and functionality of individuals with DTM pre, immediately after and 30 days of 12 treatment sessions. Method: This is a clinical trial randomised, placebo-controlled and blind, designed to study the effects of Mandibular Nonspecific Mobilization x Placebo (detuned ultrasound). Individuals will be randomised controlled trials and allocated into two groups: Group A (intervention) and Group B (placebo) and evaluated by the Research Diagnostic Criteria for Temporomandibular joint Disorders (RDC/TMD) for diagnosis of TMD, numeric scale of Pain (END), quality of life questionnaire (WHOQOL-BREF), Patient specific Functional Scale and Kinematic Analysis Tridiemsnional. Statistical Analysis: Mandibular movement will be the primary outcome and will be quantified by three-dimensional kinematic analysis. The pain, Functionality and quality of life will be the secondary outcomes. Initially the distribution of data will be checked by the Shapiro-Wilk test. In comparisons between the groups, if the data present normal distribution will be used a repeated measures ANOVA to two factors, being these: Group (intervention and placebo) and treatment (pre and post-intervention), with Bonferrone correction. If the data do not show normal distribution, a logarithmic function is used to correct striping. As level of significance will be used p < 0.05.

DETAILED DESCRIPTION:
Contextualization:Temporomandibular joint dysfunction (TMD) is defined as a group of heterogeneous changes affect a temporomandibular joint (TMJ), affecting anatomical and functional elements, is characterized as a complex and multifactorial disease. The most common signs are joint noises and limitations on the extent of the mandibular movements, associated or not to the articular disc displacement during a mandibular function and predominant symptoms are pain pre-Auricular, on ATM and/or masticatory muscles. A study of an urban brazilian population shows that 39.2% of evaluated feature at least one sign or symptom of TMD.

Its development can be related to the traumatic acometimentos of the jaw or occlusal interference or TMJ, malocclusion, changes in masticatory muscles, microtrauma caused by parafunctional habits, rheumatic diseases, emotional stress, anxiety and postural abnormalities, thus creating a major impact on quality of life and sleep of patients with this disease.

When there is a breakdown between anatomical condyle and articular eminence, disk, drift to occur for the most part, are characterized as previous joint disc displacement, with or without reduction. In both cases, the disk is presented prior to the mandibular condyle with mouth closed, and can resume his position, featuring a disc displacement with reduction (DDCR), having as main feature the snap during an opening. The disc may get introduced before the condyle during the entire opening movement, made a previous offset oral disc without reduction (DDSR), characterized by the presence of clicks, including, in the most serious cases, cause a limitation of motion and functional changes of the mandible, the adaptation of the retrodiscais tissue.

In the light of the whole complexity of the DTM it is necessary the involvement of a multidisciplinary team, including physiotherapy, with the use of manual features, have been highlighting. Manual therapy has been shown to be an important method for pain reduction, disabled and local ischemia, promoting the breakup of fibrous adhesions, improving extensibility of contractile structures, increasing range of motion. Notes that the use of Manual therapy favours the transmission of afferent information for the mecanoceptores stimulating a proprioception and a production of synovial fluid. Studies that have applied manual therapy, electing as mandibular mobilization technique in subjects with TMD, pain reduction and improvement of mandibular range. FELÍCIO et al. (2008), observed increase in WMD and pain reduction in patients treated with Orofacial Miofuncional Therapy in association with techniques such as massage therapy and a joint mobilization.

Knowledge of the movement of the jaw is important for a better understanding of the normal function of the temporomandibular joint (TMJ) and for the study of etiology, diagnosis and subsequent treatment of temporomandibular disorders. The mandibular movement also exerts influence on the joint development of the masticatory system. Therefore, knowing the three-dimensional movement of the jaw (3D) in relation to jaw is essential for clinical applications. A literature provides information on a range of motion measured by the distance between incisal edges of teeth like upper and lower incisors through digital central pachymetry and the average value of opening mouth of UM adult is approximately 50 mm. In patients with TMD buccal opening average is 32 mm and 44 mm to maximum opening without pain. In this way, pick up tools can exploit better a movement evaluation, will contribute without therapeutic success. The kinematics has been increasingly diffused in different areas of knowledge, as in gait analysis of adolescents, children, biomechanical related changes of the feet and Musculoskeletal changes related to patellofemoral syndrome, being useful also in the qualitative evaluation of the ATM graduates movements.

So, based on previous studies of our research group (AMARAL et al. 2013) (EL HAGE et al. 2013) the hypothesis of this study, on the basis of physiological changes promoted by mandibular nonspecific mobilization is a change to occur without mandibular movement and consequent reduction of signs and symptoms in patients with temporomandibular joint dysfunction.

Justification: Currently, the literature has been investigating various methods of evaluation and the possibilities of treatment of TMD. These findings highlight the current scientific clinical needs of health professionals, according to be a multifactorial origin dysfunction, with complex diagnostic and pathological mechanism which may involve several structures of the Stomatognathic system, so the more show themselves effective therapeutic resources scientifically, better treatment strategies for DTM.

Thus, this study proposes a treatment with physical therapy manual therapy technique known as Mandibular Nonspecific Mobilization, followed by the analysis of jaw movements in functional activities, carried out pre-and post-intervention physiotherapist. Their results can be of great significance and clinical trial for understanding the mandibular movement especially when the individual presents any signs and/or symptoms of TMD and there is need to perform some type of treatment and subsequent evaluation of mandibular movement. In spite of the work found in the literature with analysis of mandibular movements in patients with TMD no studies that evaluate and compare these findings after physiotherapeutic treatment, stimulating us to pick up as a manual therapy intervention can interfere with movement, through kinematic analysis.

As a result, and for reasons mentioned above, the investigators need to continue and deepen the various studies related to the treatment and evaluation of DTM (FAPESP 2013 processes/23955-6; 13/3-18354; 12/16093-5; 12/07759-0; 11/13397-0; 11/12537-3; 11/04748-4; 10/17801-8; 08/05980-5; 08/05888-1). It is known that 39.2% of the brazilian population, presents at least a sign or symptom of DTM second epidemiology study. Therefore, showing this as a national reference, and knowing that the TMD is multifactorial, the more therapeutic resources may be effective scientifically, better treatment strategies for TMD and can contribute to the public health by helping the reduction of rates of incidence, in research and in practice.

Research hypothesis: the mandibular nonspecific mobilization changes the mandibular movement and increases joint mobility in patients with TMD pre, immediately after and 30 days after 12 treatment sessions.

Null hypothesis: the mandibular nonspecific mobilization does not change the mandibular movement and does not increase joint mobility in patients with TMD pre, immediately after and 30 days after 12 treatment sessions.

General objective: The objective of this study is to evaluate the influence of mandibular nonspecific mobilization on the mandibular movement and lateralidades, in individuals with diagnosis of TMD pre, immediately after and 30 days after 12 treatment sessions.

Specific objectives: to analyse the intensity of the pain by means of numerical scale of Pain (END), immediately after and 30 days after 12 treatment sessions, analyze the quality of life through the WHOQOL-BREF questionnaire of individuals with DTM pre, immediately after and 30 days after 12 treatment sessions, analyze the functionality through the Functional Range Specifies the Patient pre, immediately after and 30 days after 12 treatment sessions.

Methodology:

It is a randomised clinical trial, placebo, controlled and blind, designed to study the effects of Mandibular Mobilization technique x Nonspecific Placebo (detuned Ultrasound). Individuals will be allocated into two groups by a randomization process in blocks (will be two blocks of 24 envelopes in total), using opaque and sealed envelopes containing: Group A = n12 (intervention) and Group B = n12 (placebo).

The evaluations will be carried out using: Research Diagnosis Criteria for Temporomandibular joint Disorders (RDC/TMD), END, WHOQOL-BREF, Functional Range Specifies the Patient, Central pachymetry and Kinematic Analysis.

The study will be divided into four phases:

Pre-intervention phase: individuals shall be recruited in accordance with the criteria for inclusion and assessed by the RDC/TMD for diagnosis of TMD. The evaluation of quality of life will be held through the WHOQOL-BREF, the intensity of the pain will be mesurada by the END, the functionality will be evaluated through Functional range Specifies the patient and mandibular movements will be captured and analyzed by Kinematic motion Analysis.

Intervention phase: individuals are randomised controlled trials in 2 groups: Group A (intervention): Mandibular Nonspecific and Mobilization Group B (placebo): using an ultrasound device detuned. The treatment will take place three times a week for 12 sessions of approximately 30 minutes each. Before and at the end of each session, the individuals will be evaluated by the END and will be held the Central pachymetry to measure the opening and lateralidades.

Post-intervention phase: in this phase will be carried out the same reviews of pre-intervention phase, which occurs immediately after the intervention phase.

Follow-up phase: one month after the last session will be held again the same pre and pos phase ratings.

Blinding: Four physiotherapists and a dentist will be part of the Protocol. One will be responsible for the evaluations. The second physical therapist will be responsible for the intervention phase, which is blind to the assessments and allocation of participants in the groups. Other physical therapist will be responsible for the performance of the kinematic analysis (a dentist will monitor the collections and will carry out the placement and removal of the brackets in the participants) and a quarter will do the processing and analysis of the data collected. The randomization and concealment of allocation will be carried out by an external developer, non-participant of the research, that will organize in opaque envelopes the individual patients and their interventions (Group A) and placebo (Group B) previously allocated. With this process, participants will have the same probability of being in one of the two treatment groups. The blinding of the evaluator and the patients will be held until the end of the research and data tabulation.

SAMPLE CALCULATION: The sample size was set from a pilot study with 8 individuals with DTM, with an average age of 28.6 ± 3.1 years and average height of 168.2 ± 10.8 cm. The average value of the oral opening movement pre (43.31 ± 5.69 mm) and post (50.83 ± 4.97) 12 sessions of mandibular nonspecific mobilization were used for this estimate. For the calculation were considered the values α = 0.05 (5% chance of type I error) and 1-β = 0.95 (% of the sample). The estimated number was of 9 individuals. Considering the possibility of a sampling of 20% loss were considered for this study 11 individuals. However, to increase the statistical power, 15 individuals per group will be used. The calculation was carried out by means of software G * Power.

STATISTICAL ANALYSIS: The mandibular movement is the primary outcome and will be for the three-dimensional kinematics analysis quantified. A pain, functionality and quality of life will be the secondary outcomes. Initially a distribution of data will be checked by the Shapiro-Wilk test. In comparisons between the groups, if the data present normal distribution is a repeated measures ANOVA notes of two factors, being these: Group (experimental and control) and treatment (pre and post-intervention), with Bonferrone correction. If the data do not show normal distribution, a logarithmic function is used to correct striping. As level of significance will be used p < 0.05. All comparisons and statistical analyses are performed using the SPSS program, version 20.0 (Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Will be included in the study, women with TMD, diagnosed by the RDC/TMD, with diversion and/or mandibular dentition full deflection (except third molars)

Exclusion Criteria:

* Not participate of the study subjects without TMD, TMD sufferers who have systemic diseases that affect the joints and/or masticatory muscles
* Over bite (bite deep) greater than 3 mm, tooth failures, neuromuscular diseases
* With hypo/condylar hyperplasia
* Making use of any type of dental prosthesis; in orthodontic treatment and/or physiotherapy
* Neurological or behavioural disorders that present that prevent the realization of kinematic analysis and/or with a history of prior surgery or orthognathic ATM.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Mandibular Movement | 45 minutes
  Mandiblulares movements will be quantified by 3D kinematics using the Vicon system ®. Markers, will be willing us participants at strategic points. The collections will be carried out before treatment, post 12 treatment sessions and follow up to a month. Static test: the volunteer will remain motionless, with his mouth shut, for 5 seconds while maintaining contact between the arches. Then a pointer is positioned in the right mandibular first Premolar and the individual in isometry is done collecting, this form will be collected the left side, upper left and right and between the upper and lower central incisors. Dynamics: will be held 6 repetitions in opening and closing freestyle to touch your teeth and will be carried out six straight tours and six excursions lefts of the mandible (laterality).

SECONDARY OUTCOMES:
WHOQOL-BREF for the evaluation of quality of life | 15 minutes
  The questionnaire is self-explanatory and can be applied in 3 ways: self administered, assisted by the interviewer or administered by the interviewer and will be applied before treatment, post 12 treatment sessions and follow up to a month.
Functional range Specifies the Patient to evaluate the functionality. | 5 minutes
  Asked to identify the patient until 3 activities that are unable to perform or presents any difficulty and may incorporate issues that were not addressed in a generic scale, but it's important for the patient's problem. The scale will be performed before treatment, post 12 treatment sessions and follow up to a month.
END to evaluate pain intensity | 5 minutes
  The degree of pain will be evaluated when an individual is at rest, before treatment, before and after each treatment session and folow up to a month.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula Amaral, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No